CLINICAL TRIAL: NCT01531946
Title: Acute MRI-techniques for the Detection of Ischemic Lesions After Transient Ischemic Attack
Brief Title: Acute MRI in Transient Ischemic Attack
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Hanne Christensen, Associate Research Professor, Consultant Neurologist, Bispebjerg Hospital
Other Study IDs: H-1-2011-75
Record Dates: First submitted 2012-02-09; First posted 2012-02-13 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Ischemic Attack, Transient
Keywords: Diffusion Tensor Imaging
MeSH Terms: conditions — Ischemic Attack, Transient | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: MRI Scan — Patients will have to spend additional 10min in the scanner.
  Additional scan modalities used:
  1. Perfusion without contrast: Arterial spin labeling (ASL) with the ability of showing signs of ischemia.
  2. Diffusion tensor imaging (DTI): Has a higher sensitivity than DWI in displaying local ischemic lesions.
  An overall 20min scan period.

SUMMARY:
The purpose of this study is to detect acute ischemic lesions in patients admitted with symptoms of transient ischemic attack (TIA).

Diffusion weighted Imaging (DWI) is today one of the best ways to detect ischemic lesions after TIA. The problem is that this only gives the diagnosis in 30% of the cases.

It is possible that the addition of Arterial spin labeling (ASL) perfusion imaging and diffusion tensor imaging will make it possible to give a more accurate diagnosis.

DETAILED DESCRIPTION:
The purpose of this study is to detect acute ischemic lesions in patients admitted with symptoms of transient ischemic attack (TIA).

Diffusion weighted Imaging (DWI) is today one of the best ways to detect ischemic lesions after TIA. The problem is that this only gives the diagnosis in 30% of the cases.

It is possible that the addition of ASL-perfusion imaging and diffusion tensor imaging will make it possible to give a more accurate and selective diagnosis of TIA.

Patients admitted with clinical signs of TIA can be included. Patients will be examined with the TIA protocol in reference to the standardized clinical care:

1. 1,5 tesla gradient echo and 3 tesla Susceptibility weighted imaging (SWI) to detect microbleed as sign of small vessel disease.
2. Axial T2 FLAIR to detect white matter lesions.
3. Axial DWI to detect areas with impeded diffusion.

(Total scantime 10min)

If no signs of ischemic lesions is detected the following additional research scan-protocol will be initiated:

1. Perfusion without contrast: Arterial spin labeling (ASL) with the ability of showing signs of ischemia.
2. Diffusion tensor imaging (DTI): Has a higher sensitivity than DWI in displaying local ischemic lesions.

(Total additional scantime 10min)

All in All 20min in the scanner.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of TIA
* Informed consent
* No serious respiratory or cardiac implications

Exclusion Criteria:

* Contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the stroke ward at Bispebjerg University Hospital with signs of TIA.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2012-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
frequency of patients with ischaemic lessions on DTI | on first MRI
  We want to assess the frequency of patients in whom a diffusion restricted lesion can only be observed on DTI

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Christensen, MD, DMSci, Principal Investigator — Department of Neurology and Cerebrovascular Diseases, Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Background] Luengo-Fernandez R, Gray AM, Rothwell PM. Effect of urgent treatment for transient ischaemic attack and minor stroke on disability and hospital costs (EXPRESS study): a prospective population-based sequential comparison. Lancet Neurol. 2009 Mar;8(3):235-43. doi: 10.1016/S1474-4422(09)70019-5. Epub 2009 Feb 4. PMID 19200786
- [Background] Olivot JM, Albers GW. Diffusion-perfusion MRI for triaging transient ischemic attack and acute cerebrovascular syndromes. Curr Opin Neurol. 2011 Feb;24(1):44-9. doi: 10.1097/WCO.0b013e328341f8a5. PMID 21157338
- [Background] Schaefer PW, Copen WA, Lev MH, Gonzalez RG. Diffusion-weighted imaging in acute stroke. Magn Reson Imaging Clin N Am. 2006 May;14(2):141-68. doi: 10.1016/j.mric.2006.06.005. PMID 16873008
- [Derived] Havsteen I, Willer L, Ovesen C, Nybing JD, AEgidius K, Marstrand J, Meden P, Rosenbaum S, Folke MN, Christensen H, Christensen A. Significance of arterial spin labeling perfusion and susceptibility weighted imaging changes in patients with transient ischemic attack: a prospective cohort study. BMC Med Imaging. 2018 Aug 20;18(1):24. doi: 10.1186/s12880-018-0264-6. PMID 30126352
- [Derived] Havsteen I, Ovesen C, Willer L, Nybing JD, AEgidius K, Marstrand J, Meden P, Rosenbaum S, Folke MN, Christensen H, Christensen A. Small cortical grey matter lesions show no persistent infarction in transient ischaemic attack? A prospective cohort study. BMJ Open. 2018 Jan 21;8(1):e018160. doi: 10.1136/bmjopen-2017-018160. PMID 29358426
- [Derived] Havsteen I, Ovesen C, Willer L, Nybing JD, AEgidius K, Marstrand J, Meden P, Rosenbaum S, Folke MN, Christensen H, Christensen A. Comparison of 3- and 20-Gradient Direction Diffusion-Weighted Imaging in a Clinical Subacute Cohort of Patients with Transient Ischemic Attack: Application of Standard Vendor Protocols for Lesion Detection and Final Infarct Size Projection. Front Neurol. 2017 Dec 18;8:691. doi: 10.3389/fneur.2017.00691. eCollection 2017. PMID 29326651